CLINICAL TRIAL: NCT05124470
Title: Pilot Study Evaluating the Feasibility and the Preliminary Effects of a Cognitive Remediation Method by Rhythmic, Vocal and Embodied Musical Learning for Stabilized Schizophrenic Patients.
Brief Title: Cognitive Remediation Method by Rhythmic, Vocal and Embodied Musical Learning for Stabilized Schizophrenic Patients
Acronym: ARCoS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/20/0448
Record Dates: First submitted 2021-10-27; First posted 2021-11-18 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia
Keywords: Psychiatric Rehabilitation; Music Therapy; Cognitive Remediation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- musical training sessions (Experimental): 24 musical training sessions over the 6 months + 3 months of follow-up post cognitive remediation.
  Interventions: Other: cognitive remediation by musical training sessions

INTERVENTIONS:
Other: cognitive remediation by musical training sessions — The musical learning method "Diapason & Metronome" is unprecedented. It was specially created by Florent Cholat. It aims an apprenticeship of a musical practice adapted to subjects with schizophrenia. The method does not require the handling of a musical instrument; it is based on the voice and the body. It is built on the three essential dimensions of music, which are rhythm, single sound and harmony. "Rhythm" concerns the division and management of time. The "single sound" allows work on the representation of a sound object as a singularity. "Harmony" allows you to work on the positioning of a sound in the globality of the chord to which it belongs and in the collective polyphony exercises.

SUMMARY:
ARCoS is a pilot study evaluating the feasibility and preliminary effects of a method of cognitive remediation by a Rhythmic, Vocal and Embodied Musical Learning for a population of stabilized schizophrenic patients. 20 stabilized schizophrenics patients will participate in the study for 9 months, i) 6 months of Musical learning (24 sessions over the 6 months) ; ii) and 3 months of follow-up post cognitive remediation. Assessments of attention deficits, inhibitory abilities, negative symptoms and anxiety, will carried out at baseline (V1, M0), third month (M3), sixth month (M6) after the start of the intervention and third months after the end of the intervention (M9).

The primary endpoint will be the proportion of patients who have attended at least 80% of the musical training sessions over the 6 months (participation in at least 19/24 sessions).

DETAILED DESCRIPTION:
Schizophrenia is a chronic psychiatric condition affecting 1% of the population. Antipsychotic medications are effective on positive symptoms (delusions, hallucinations). However, they do not have a significant effect on negative symptoms (apragmatism, social withdrawal, blunting of affect, etc.) and cognitive impairment. These last two dimensions are the most impacting in terms of social functioning and quality of life, and antipsychotics can potentially aggravate them. In addition to pharmacological treatments it is recommended to combine non-pharmacological approaches including cognitive remediation and psychosocial rehabilitation. The latter are best able to improve the personal and interpersonal functioning of patients and improve their quality of life which makes a recovery trajectory possible. Do date very few studies conduct cognitive remediation using musical learning. We have created an original teaching method based on the embodied dimension of cognition.

The objective is to conduct a first pilot study to validate the feasibility of this music learning with schizophrenic patients. It will allow a preliminary evaluation of the effects of this new approach on cognitive disorders and negative symptoms of stabilized schizophrenic patients.

20 stabilized schizophrenics patients will participate in the study for 9 months, i) Rhythmic, Vocal and Embodied Musical Learning to two groups of 10 patients during 6 months each. (24 sessions over the 6 months) ; ii) and 3 months of follow-up post cognitive remediation. Each patient will have 4 evaluation visits during the study.

ELIGIBILITY:
* Inclusion criteria:

  1. Established schizophrenia or with schizoaffective disorder as per Diagnostic and Statistical Manual (DSM 5)
  2. Clinically stable (with no full-time hospitalization within the last 6 months)
  3. Regular follow-up (followed in a day Hospital of Psychiatric)
  4. Patient must be on stable background antipsychotic treatment (with no modification within the last 6 month)

  4. Male or female patients who are 18-60 years of age 5. Signed and dated written consent 6. Patient having a health Insurance coverage
* Exclusion criteria:

  1. Patient with moderate to severe intellectual disabilities (clinical criteria)
  2. Addictive comorbidity (excluding tobacco and behavioral addictions)
  3. Previous neurologic pathology with cognitive impact
  4. Patient who are following a cognitive rehabilitation program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
proportion of patients who have attended at least 80% of the musical training sessions over the 6 months | 6 months
  The primary outcomes will be the proportion of patients who have attended at least 80% of the musical training sessions over the 6 months (participation in at least 19/24 sessions).

SECONDARY OUTCOMES:
list of factors of no adherence to musical learning | 6 months
  Describe the causes of no adherence to the project and the difficulties encountered during the study.
Reduce of attention deficits at 6 month | 6 months
  change of score of attention deficit (d2-R : Revised Focused Attention Test) between inclusion and the end of the program (M6)
Reduce of attention deficits at 9 month | 9 months
  change of score of attention deficit (d2-R : Revised Focused Attention Test) between inclusion and 3 months after (M9)
Improving inhibitory abilities at 6 month | 6 months
  change of score of attention deficit (Go-no-Go) between inclusion and the end of the program (M6)
Improving inhibitory abilities at 9 month | 9 months
  change of score of attention deficit (Go-no-Go) between inclusion and 3 months after (M9)
Decrease on Negative symptoms | 6 months
  change of score the Self evaluation of negative symptoms (SNS) between inclusion and the end of the program (M6), and between inclusion and 3 months after (M9)
The state of anxiety at 6 month | 6 months
  change of scores of State-Trait Anxiety Inventory (STAI) between inclusion and the end of the program (M6)
The state of anxiety at 9 month | 6 months
  change of scores of State-Trait Anxiety Inventory (STAI) between inclusion and 3 months after (M9)
modification of psychotropic medication | 6 months
  The modification of psychotropic medication at the end of the program compared to inclusion
modification of psychotropic medication | 9 months
  The modification of psychotropic medication at 3 months after (post cognitive remediation phase) compared to inclusion

CONTACTS AND LOCATIONS:
Overall Officials: TUDI L GOZE, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - CH Marchant, Toulouse
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No